CLINICAL TRIAL: NCT06926127
Title: Genomic Profiling of GENetic & RARE Diseases for the Customization of Care and Prevention Pathways
Brief Title: Genomic Profiling of Genetic and Rare Diseases
Acronym: GEN&RARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6987
Record Dates: First submitted 2024-10-11; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-10

CONDITIONS: Rare Diseases; Genetic Disease
MeSH Terms: conditions — Rare Diseases; Genetic Diseases, Inborn | interventions — Exome Sequencing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients with suspected rare or specific genetic diseases diagnosed based on clinical presentation and instrumental examination performed by geneticist or by a specialist physician experienced in the specific condition (e.g., phenotype associated with a known genetic syndrome, known neuromuscular disease, or known specific regional disease such as hypertrophic/dilated cardiomyopathy) are enrolled to undergo genetic testing for diagnostic purposes and to improve personalized treatment.
  Interventions: Genetic: Whole Exome Sequencing (WES)

INTERVENTIONS:
Genetic: Whole Exome Sequencing (WES) — Blood samples, buccal swabs, and pathological tissue samples (skin/muscle) will be collected, and subsequently, DNA extracted from those tissues will be used for genomic analysis using Whole Exome Sequencing. The sample will follow the diagnostic pipeline already established inside the hospital. Moreover, the remaning aliquots of DNA extracted from the tissue (peripheral blood or tissue specimen) will be sent by the Genomics core facility to the Biobank for storage upon analysis completion.

SUMMARY:
In Italy, over 2 million patients are affected by Rare Diseases (RD), which pose significant challenges due to their clinical diversity, long diagnostic processes (often 4-5 years), and high socio-healthcare costs. The Italian healthcare system has recognized these challenges, leading to initiatives like a national Rare Diseases (RD) registry, a comprehensive list of Rare Diseases (RDs) eligible for healthcare exemptions, and the establishment of a National Committee for Rare Diseases. Research on the genetic mechanisms of Rare Diseases (RDs) is robust, particularly for innovative therapies, and ranks second to oncology.

The Policlinico Universitario A. Gemelli IRCCS Foundation serves as a key reference institute for Rare Diseases (RD) in Lazio, managing over 10,000 patients through accredited centers. A recent initiative aims to enhance the Rare Diseases network by integrating genomic knowledge with clinical practice. The project focuses on utilizing Next Generation Sequencing (NGS) for early genetic diagnosis, promoting personalized medicine.

Given the challenges the National Health Service faces in resource allocation for Rare Diseases (RD) and the recent approval of a new outpatient healthcare tariff, this initiative is timely. The foundation seeks to replace targeted genetic tests with Whole Exome Sequencing (WES), increasing the identification of molecular conditions and reducing diagnostic turnaround times.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-90 years
* Patients with suspected rare disease/genetic disease diagnosed based on the clinical criteria/instrumental examination performed by a reference physician experienced in the specific condition (e.g., phenotype attributable to a known genetic syndrome, known neuromuscular disease, known organ-specific disease such as hypertrophic/dilated cardiomyopathy) to undergo genetic analysis
* Patients with a phenotype suggestive of a rare disease/genetic disease not specifically linked to a known condition
* Patients with suspected rare disease/genetic disease, who have undergone quantitative genetic analyses (e.g., array-CGH) or qualitative analyses (e.g., NGS panel of known genes), which yielded negative results
* Patients who have already received a genetic etiological diagnosis and for whom the current project can address further questions such as the personalization of a prevention or therapy pathway.

Exclusion Criteria:

* Individuals (patients, parents, and/or legal guardians) who refuse to participate in the project for any reason.

Ages: 1 Minute to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Reduce diagnostic timelapse of rare genetic conditions | from 1 year to 4 years
  To reduce the time frame between first clinical evaluation to molecular diagnosis by improve the genomic characterization of rare genetic conditions trought implementation of the actual molecular analysis (from targeted panels to whole exome sequencing - WES

SECONDARY OUTCOMES:
Improve the hospital's diagnostic rate | 5 years
  Improving the hospital's diagnostic rate by evaluating data collected from the analysis of 1500 biological samples with the Illumina Novaseq 6000 exome sequencing system.
Identify an increasing number of molecular variants | 5 years
  Identify an increasing number of disease causing genes in rare conditions on 1500 biological samples processed with the Illumina Novaseq 6000 exome sequencing system.
Reduce healthcare costs for a definitive diagnosis | 5 years
  Reduce costs for molecular analysis to reach a definitive diagnosis by using untargeted molecular test (WES) vs multiple targeted panels often needed for complex rare disesases

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC PEDIATRIA, Rome, Lazio, Italy